CLINICAL TRIAL: NCT00324090
Title: Glycemic Index, Body Weight and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danone Vitapole, France. (Unknown); Masterfoods Denmark (Other); Euryza GmbH, Germany. (Unknown); Cerealia R&D, Schulstad Brød A/S, Denmark. (Unknown); Lund University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: (KF) 01-249/01; B184
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2002-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

INTERVENTIONS:
Behavioral: High and low glycemic index

SUMMARY:
The purpose of this study is to investigate the effect of a diet with either high or low glycemic index (GI) on ad libitum (free) food intake, body weight, fat mass and fat-free mass, risk markers for diabetes and cardiovascular diseases, energy expenditure and substrate oxidation after 10 weeks´ intake in slightly overweight subjects.

DETAILED DESCRIPTION:
Experimental design Two matched groups are given high-GI or low-GI foods to their own diet throughout 10 weeks in a parallel design. A number of measurements are done before, during and at the end of the 10 weeks' intervention.

Subjects A total of 50 slightly overweight (body mass index, BMI = 25-30 kg/m2) women, 20-40 years of age participate. Subjects are randomized according to body weight, composition, age, sex and physical activity level into two matched groups.

A representative subgroup of 15 subjects is randomized from each diet group (a total of 30 subjects) for measurements of energy expenditure and substrate oxidation by ventilated hood as well as postprandial blood sampling.

Experimental diets Subjects eat their own diet until the intervention starts and perform a 7-day weighed dietary record for determination of habitual food intake. At the beginning and every 2 weeks during the 10 weeks' intervention all subjects are instructed in consuming a low-fat (<30 E%), high-carbohydrate diet (>55 E%) by a dietician. Subjects are each week given an amount of carbohydrate-rich foods with either high or low GI with instructions to consume a minimum amount of these every day. We aim at controlling about 75% of the subjects' total carbohydrate intake. The exact amount of test foods eaten is noted every day by the subjects by use of a diary and a diet scale. Instructions in food intake and cooking recipes are given by the dietician. A positive list and a negative list of food items is provided for each study group.

Besides the fixed minimum amount of experimental foods subjects can eat at liberty. Another 7-d dietary record is performed at week 5 and week 10 to register ad libitum food intake. To further validate the dietary records 24-h urine samples are taken during the registrations. Lithium will also be added to the experimental foods in week 4-5 to follow compliance during the study.

Measurements

All subjects:

Week 0, 2, 4, 6, 8, 10 we measured body weight,fat mass and fat-free mass using bio-electrical impedance.In week 0 and 10 we measured body composition by DEXA-scan, W/H-ratio and sagittal height. Blood samples fasting in week 0 and 10 (Glucose, insulin, triacylglycerol (TAG), non-esterified fatty acids (NEFA), leptin, T-cholesterol, LDL-chol, HDL-chol, fructosamine, glycated hemoglobin, GIP, GLP-1, GLP-2, ghrelin, factor VIIc, factor VIIb, PAI-1, Apo A IV.). Blood pressure in week 0 and 10 (fasting systolic and diastolic BP and heart rate). 24-h urine sample is collected in week 0, 5 and 10. Feces is collected in the subgroup in week 0 and 10.

Subgroup:

Week 10: Ventilated hood for measurement of fasting and 4-h postprandial energy expenditure and substrate oxidation. Postprandial appetite scores for hunger, satiety, fullness, prospective consumption, desire for something sweet, fatty. Postprandial blood samples for 4 hours after breakfast (30, 60, 90, 120, 180, 240 min): Glucose, insulin, NEFA, TAG, leptin, glucagon, GIP, GLP-1, GLP-2, ghrelin, paracetamol. At 240 min: factor VIIbt, PAI-1, Apo A IV.

ELIGIBILITY:
Inclusion Criteria:

* healthy, slightly overweight (body mass index, BMI = 25-30 kg/m2) women, premenopausal, non-alcoholic (< 14 units alcohol/w)

Exclusion Criteria:

* smoking, elite athletes, food allergies, pregnant, lactating, on medication, blood donation 3 months before, during and 3 months after the completion of the study

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43
Dates: Start 2002-03; Study Completion 2002-07

PRIMARY OUTCOMES:
Body weight
Fat mass and fat-free mass
Food intake

SECONDARY OUTCOMES:
Risk markers for diabetes and CVD
Energy expenditure and substrate oxidation
Appetite

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Prof, Principal Investigator — Department of Human Nutrition, Centre for Advanced Food Studies, The Royal Veterinary and Agricultural University, Denmark

REFERENCES:
- [Derived] Krog-Mikkelsen I, Sloth B, Dimitrov D, Tetens I, Bjorck I, Flint A, Holst JJ, Astrup A, Elmstahl H, Raben A. A low glycemic index diet does not affect postprandial energy metabolism but decreases postprandial insulinemia and increases fullness ratings in healthy women. J Nutr. 2011 Sep;141(9):1679-84. doi: 10.3945/jn.110.134627. Epub 2011 Jul 20. PMID 21775528
- [Derived] Jensen L, Sloth B, Krog-Mikkelsen I, Flint A, Raben A, Tholstrup T, Brunner N, Astrup A. A low-glycemic-index diet reduces plasma plasminogen activator inhibitor-1 activity, but not tissue inhibitor of proteinases-1 or plasminogen activator inhibitor-1 protein, in overweight women. Am J Clin Nutr. 2008 Jan;87(1):97-105. doi: 10.1093/ajcn/87.1.97. PMID 18175742